CLINICAL TRIAL: NCT01463930
Title: Effects of an Educational Audiovisual Videodisc on Patients' Pre-operative Expectations With Total Knee Replacement: a Randomized Study
Brief Title: Audiovisual Videodisc Education and Modification of Expectations With Total Knee Replacement (TKR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Joan Leal Blanquet, MD, MSc, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PSMARCOT01_2011
Record Dates: First submitted 2011-10-16; First posted 2011-11-02 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Total Knee Replacement
Keywords: Total Knee Replacement; Expectations; Audiovisual videodisc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Audiovisual videodisc and medical verbal information (Experimental)
  Interventions: Behavioral: Educational audiovisual videodisc and medical verbal information
- Medical verbal information (Active Comparator)
  Interventions: Behavioral: Medical verbal information

INTERVENTIONS:
Behavioral: Educational audiovisual videodisc and medical verbal information — General and specific medical verbal information and ten-minute DVD where the process from admission to the surgical intervention, recovery room, immediate postoperative care, and outpatient care at two, six, and twelve months after surgery was shown. The video included experiences of patients with respect to pain and function and examples of functionality during daily life activities such as stairs, kneeling or squatting. The video also demonstrated the facilities and rehabilitation techniques employed in the Physical Medicine and Rehabilitation Service.
  Arms: Audiovisual videodisc and medical verbal information
Behavioral: Medical verbal information — General and specific verbal information provided by both the surgeon and a specialized nurse including basics of surgical technique, potential complications, and rehabilitation.
  Arms: Medical verbal information

SUMMARY:
Information provided to patients modifies their expectations with surgery. The effects of preoperative audiovisual information on expectations with total knee replacement (TKR) have not been investigated. The purposes of this study were to investigate the effectiveness of an educational videodisc on the modification of pre-operative patients' expectations with TKR and to find a biophysical profile of subjects in whom this videodisc could be most effective. It was hypothesized that patients receiving standard information plus additional medical information through audiovisual videodiscs would modify their pre-operative expectations more than those only receiving the standard information through medical interviews.

ELIGIBILITY:
Inclusion Criteria:

* Patients with knee osteoarthritis waiting for total knee replacement.

Exclusion Criteria:

* Cognitive disorders or language barriers precluding medical interview.
* Contralateral total knee replacement.
* History of revision total knee replacement.
* History of unicompartmental knee arthroplasty

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in patient-reported postoperative expectatives about the results of total knee replacement to inmediately after receiving audiovisual plus verbal information (intervention grou) or only verbal information (control group) | Baseline and 1 month later (1 month before surgery)
  The study measures the patient's expectatives about the improvement of pain, function, and psychological well-being after undergoing total knee replacement. These expectatives are measured through the Hospital for Special Surgery Knee Replacement Expectations Survey (KRES), and a score ranging from 0 to 100 is reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de l'Esperança - Parc de Salut MAR, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Mancuso CA, Sculco TP, Wickiewicz TL, Jones EC, Robbins L, Warren RF, Williams-Russo P. Patients' expectations of knee surgery. J Bone Joint Surg Am. 2001 Jul;83(7):1005-12. doi: 10.2106/00004623-200107000-00005. PMID 11451969
- [Background] Noble PC, Conditt MA, Cook KF, Mathis KB. The John Insall Award: Patient expectations affect satisfaction with total knee arthroplasty. Clin Orthop Relat Res. 2006 Nov;452:35-43. doi: 10.1097/01.blo.0000238825.63648.1e. PMID 16967035
- [Background] Hepinstall MS, Rutledge JR, Bornstein LJ, Mazumdar M, Westrich GH. Factors that impact expectations before total knee arthroplasty. J Arthroplasty. 2011 Sep;26(6):870-6. doi: 10.1016/j.arth.2010.09.010. Epub 2010 Nov 12. PMID 21074356
- [Background] Mancuso CA, Salvati EA, Johanson NA, Peterson MG, Charlson ME. Patients' expectations and satisfaction with total hip arthroplasty. J Arthroplasty. 1997 Jun;12(4):387-96. doi: 10.1016/s0883-5403(97)90194-7. PMID 9195314
- [Background] Nilsdotter AK, Toksvig-Larsen S, Roos EM. Knee arthroplasty: are patients' expectations fulfilled? A prospective study of pain and function in 102 patients with 5-year follow-up. Acta Orthop. 2009 Feb;80(1):55-61. doi: 10.1080/17453670902805007. PMID 19234886